CLINICAL TRIAL: NCT06855706
Title: Life on the Go 3: A Randomized Controlled Trial of Automated, Personalized Physical Activity Intervention Using Wearable Devices to Improve Immune Function and Clinical Outcomes in Ovarian and Endometrial Cancer Patients
Brief Title: An Automated Personalized Physical Activity Intervention to Improve Immune Function and Clinical Outcomes in Stage II-IV Ovarian, Primary Peritoneal or Fallopian Tube Cancer and Newly Diagnosed Endometrial Cancer, Life on the Go 3 Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 4260824; NCI-2025-00835 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 4260824 (Other: Roswell Park Cancer Institute); P50CA159981 (NIH)
Record Dates: First submitted 2025-02-20; First posted 2025-03-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Stage II Fallopian Tube Cancer AJCC v8; Stage II Ovarian Cancer AJCC v8; Stage II Primary Peritoneal Cancer AJCC v8; Stage III Fallopian Tube Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Primary Peritoneal Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8
MeSH Terms: conditions — Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Behavior Therapy; Practice Guidelines as Topic; Standard of Care; Specimen Handling; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Personalized Physical Activity intervention) (Experimental): Patients receive personalized PA goals and positive feedback to increase participation in MVPA in 10-15 minute increments up to 150 minutes per week for 12 weeks then sustain participation for an additional 12 weeks (6 months total). Patients also receive ongoing support to maintain or further increase PA levels up to month 6. Patients wear a Fitbit Sense 2 and CGM device continuously throughout the 6 month intervention. Additionally, patients undergo blood sample collection throughout the study.
  Interventions: Behavioral: Behavioral Intervention; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Exercise Intervention; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Supportive Care
- Arm II (Standard PA) (Active Comparator): Patients receive general PA counseling recommending 150 minutes of activity per week consistent with standard of care at time of enrollment. Patients also wear a Fitbit Sense 2 and CGM device for 6 months. Additionally, patients undergo blood sample collection throughout the study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Receive personalized PA goals and positive feedback
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (Personalized Physical Activity intervention)
Other: Best Practice — Receive general PA counseling
  Other Names: standard of care; standard therapy
  Arms: Arm II (Standard PA)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Ancillary studies
Other: Exercise Intervention — Participate in MVPA
  Arms: Arm I (Personalized Physical Activity intervention)
Other: Medical Device Usage and Evaluation — Wear a Fitbit Sense 2 and CGM device
Other: Questionnaire Administration — Ancillary studies
Other: Supportive Care — Receive ongoing support
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Arm I (Personalized Physical Activity intervention)

SUMMARY:
This clinical trial compares the effect of an automated personalized physical activity intervention supported by wearable technology to standard of care on physical activity levels and quality of life in patients with stage II- IV ovarian, primary peritoneal, fallopian tube cancer or endometrial cancer that is newly diagnosed. Physical activity is a modifiable risk factor for the prevention and treatment of many diseases. In fact, increased levels of physical activity have been shown to decrease the risk of some cancers as well as increase overall survival in some cancers. Currently, standard of care guidelines include participation in at least 150 minutes of moderate exercise weekly. An automated personalized physical activity intervention may increase physical activity, enhance quality of life, and improve physical function and daily living activities compared to standard recommendations in patients with stage II-IV ovarian, primary peritoneal, fallopian tube or newly diagnosed endometrial cancer. This trial also evaluates the impact of physical activity on the gut microbiome and immune function. The microbiome is the collection of tiny organisms, like bacteria, that live in and on the body, especially places like the gut. These microorganisms play an important role in health. Information gathered from this study may help understand how the gut microbiome and physical activity influences the immune system in patients with stage II-IV ovarian, primary peritoneal, fallopian tube or newly diagnosed endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether an automated, personalized physical activity (PA) intervention using wearable technology increases the proportion of patients with ovarian or endometrial cancer who achieve at least 150 minutes of moderate to vigorous physical activity (MVPA) per week by the end of the first 3 months, compared to standard recommendations.

SECONDARY OBJECTIVES:

I. To assess whether the physical activity (PA) intervention leads to sustained increases in physical activity levels among patients with ovarian or endometrial cancer by measuring the proportion of participants who maintain at least 150 minutes of moderate to vigorous physical activity (MVPA) per week on average during the last three months of the intervention period (months 4 to 6).

II. To evaluate changes in average weekly active minutes from baseline to 3 months and 6 months between the intervention and control groups.

III. To evaluate the effect of the PA intervention on quality of life among ovarian and endometrial cancer patients, as measured by validated questionnaires.

IV. To assess changes in physical functioning and activities of daily living between the intervention and control groups.

OUTLINE: Patients are randomized to 1 of 2 groups.

ARM I: (PA INTERVENTION): Patients receive personalized PA goals and positive feedback to increase participation in MVPA in 10-15 minute increments up to 150 minutes per week for 12 weeks then sustain participation for an additional 12 weeks (6 months total). Patients also receive ongoing support to maintain or further increase PA levels up to month 6. Patients wear a Fitbit Sense 2 and CGM device continuously throughout the 6 month intervention. Additionally, patients undergo blood sample collection throughout the study.

ARM II (STANDARD PA): Patients receive general PA counseling recommending 150 minutes of activity per week consistent with standard of care at time of enrollment. Patients also wear a Fitbit and continuous glucose monitor (CGM) device for 6 months. Additionally, patients undergo blood sample collection throughout the study.

After completion of study intervention, patients are followed up every 3 months for up to 24 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old on day of signing informed consent
* Have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Participant must satisfy one of the following conditions:

  * Have a clinically suspected or confirmed diagnosis of stage II-IV ovarian, primary peritoneal, or fallopian tube cancer by clinical presentation and elevated CA-125 and may be awaiting staging surgery or tumor tissue biopsy followed by neoadjuvant chemotherapy. Inclusion of clinically suspected ovarian cancer cases is because we want to capture data starting from the earliest point of the diagnostic pathway and before definitive staging surgery. This allows us to assess the impact of physical activity and the feasibility of wearable device monitoring as patients transition into neoadjuvant chemotherapy and potential surgery
  * Have recurrent ovarian, primary peritoneal, or fallopian tube cancer at any time point of their recurrence, if they meet eligibility criteria (any histology accepted). Inclusion of recurrent ovarian cancer cases is because ovarian cancer often recurs, and understanding physical activity patterns and interventions in patients experiencing recurrence is critical for comprehensive insights. This ensures the study includes the continuum of disease management beyond initial diagnosis
  * Have pre-operative biopsy-proven endometrial cancer (endometrioid, serous, mucinous, or clear cell, poorly differentiated) with plans for surgical resection using a minimally invasive approach or medical management with chemotherapy combination, hormonal treatment or radiation. Inclusion of biopsy-proven endometrial cancer cases but not clinically suspected or recurrent cases is because we are focusing on confirmed, newly diagnosed patients who will undergo surgical resection or medical management
* willing to wear the activity tracking device for at least 70% of their waking hours each day (11 hours/day) throughout the 6-month study period
* under the care of Roswell Park Comprehensive Cancer Center during the study period, which includes one or more of the following:

  * Receiving cancer treatment at Roswell Park Comprehensive Cancer Center
  * Undergoing surgery at Roswell Park Comprehensive Cancer Center
  * Participating in surveillance visits at Roswell Park Comprehensive Cancer Center
  * Receiving adjuvant treatment at an outside facility but returning to Roswell Park Comprehensive Cancer Center for periodic consultation visits and agreeing to comply with all study procedures, including data sharing from external providers
* willing to participate in questionnaires and blood and stool collection throughout the study for translational research purposes
* Participant must understand the investigational nature of this study and sign an independent ethics committee/institutional review board approved written informed consent form prior to receiving any study related procedure
* Have a smartphone with daily internet access that is compatible with the wearable devices and applications used in the study (e.g., Fitbit Sense 2 and CGM applications)

  * NOTE: Patients who are already achieving or exceeding the goal of 150 minutes of physical activity per week are eligible for this study. This inclusion is intentional, as the study aims to evaluate the full spectrum of physical activity levels-both baseline activity and changes over time-and their relationship with clinical outcomes, metabolic measures (e.g., glucose levels), inflammation, and physical function

Exclusion Criteria:

* serious psychiatric illness that is not currently stabilized, including but not limited to:

  * Schizophrenia or other psychotic disorders
  * Bipolar disorder
  * Sever major depressive disorder
  * Severe personality disorders diagnosed by a qualified mental health professional
  * Recent suicide attempt or psychiatric hospitalization within the previous 12 months
* Life expectancy of less than 12 months, as determined by the Investigator based on clinical judgment and available prognostic tools
* history of other invasive malignancies within the last two years, except for:

  * Non-melanoma skin cancer
  * In situ cervical cancer
* resting heart rate greater than 120 beats per minute after 10 minutes of seated rest, confirmed on two separate measurements
* systolic blood pressure greater than 180 mmHg or diastolic blood pressure greater than 100 mmHg, measured after 10 minutes of seated rest, confirmed on two separate measurements
* Unstable angina or myocardial infarction within the past 3 months.

  * Unstable Angina: Chest pain at rest or chest pain of increasing frequency, severity, or duration that requires medical attention
  * Myocardial Infarction: Heart attack diagnosed by a medical professional
* Pregnant or nursing participants will be excluded, as confirmed via urine test during screening procedures.
* unwilling or unable to follow the protocol requirements, including but not limited to:

  * Cognitive impairment that affects the ability to provide informed consent or comply with study procedures
  * Language barriers without access to adequate translation services
  * Lack of access to necessary technology (e.g., smartphones compatible with study devices)
  * Other factors that would prevent adherence to study protocols
* Any condition which, in the Investigator's opinion, makes the patient unsuitable for participation in the study or may interfere with the patient's ability to comply with the study requirements or the safety of the patient. Conditions may include, but are not limited to:

  * Severe pulmonary disease
  * Uncontrolled metabolic disorders
  * Other significant medical conditions that pose a risk during increased physical activity
* Participants who do not provide a valid cell phone number or do not consent to receive SMS messages from Fitabase for motivational and compliance monitoring purposes will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving ≥ 150 minutes of moderate to vigorous physical activity (MVPA) per week | At 3 months (weeks 11 and 12)
  Will be defined based on Fitbit's activity intensity levels (e.g., minutes spent in moderate and vigorous zones). Fisher's exact test will be used to compare proportions between groups. Will use logistic regression for adjustments for baseline physical activity levels if necessary. A two-sided alpha = 0.05 will be used for statistical significance.

SECONDARY OUTCOMES:
Proportion of participants maintaining ≥150 minutes of MVPA per week on average | During months 4-6 (weeks 13-24) of the intervention period
  MVPA will be based on Fitbit's activity intensity levels (e.g., minutes spent in moderate and vigorous zones). Will be compared between groups using the Fisher's exact test.
Mean change in average weekly active minutes | From baseline to 3 and 6 months
  Mean changes in average weekly active minutes will be calculated within and between groups. Linear mixed-effects models will be used to assess changes over time between groups and adjusted for baseline activity levels and other covariates.
Changes in quality of life (QOL) scores -Ovarian Cancer Module | From baseline to 3 and 6 months
  Will be evaluated using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)- Ovarian (OV)28 . The difference in mean change of QOL scores between the intervention and control groups will be analyzed using analysis of covariance (ANCOVA), adjusting for baseline scores. 28 questions rated on a 4 point rating scale : "Not at all," "A little," "Quite a bit," and "Very much."
Changes in Quality of life | From baseline to 3 and 6 months
  36-item Short form Survey (SF-36)Patient-reported outcome measurement for health-related quality of life and activities of daily living scored on a scale of 0 (negative health) to 100 (positive health).
Change in Quality of Life Score- Endometrial | From baseline to 3 and 6 months
  EORTC QLQ - Endometrial (EN) 24.he EORTC QLQ-EN24 is a 24-item instrument designed to assess various aspects of treatment-related quality of life specifically in patients undergoing treatment for endometrial cancer.The EORTC QLQ-EN24 uses a 4-point response scale for most items: 1 = not at all, 2 = a little, 3 = quite a bit, and 4 = very much.
  A higher score indicates worse quality of life.
Functional Status | From baseline to 3 and 6 months
  Will compare difference in mean change of Lawton Instrumental Activities of Daily Living Scale (IADL) . Statistical analysis will use paired t-tests or non-parametric equivalents if data are not normally distributed. Changes will be analyzed using ANCOVA. Non-parametric tests may be used if data are not normally distributed.
Functional Status - Katz Index of Activities Daily Living | From baseline to 3 and 6 months
  Activities of daily living as assessed by the KATz Index. A score of 6 is high whereas a score of 0 is low.

CONTACTS AND LOCATIONS:
Overall Officials: Emese Zsiros, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States